CLINICAL TRIAL: NCT04388618
Title: Investigating Anosmia and Ageusia in COVID-19 Adult Patients in Saudi Arabia
Status: Completed | Type: Observational
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, osama y kentab, m.d, FAAP, FACEP , CLINICAL ASSOCIATE PROFESSOR OF EMERGENCY MEDICINE, SENIOR CONSULTANT PEDIATRIC EMERGENCY MEDICINE, Princess Nourah Bint Abdulrahman University
Other Study IDs: H-01-R-059
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Anosmia; Ageusia; Covid19; Corona Virus Infection
Keywords: anosmia; ageusia; covid19; corona virus infection
MeSH Terms: conditions — Anosmia; Ageusia; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid19 positive patients: participants who present with signs and symptoms suspected for covid19 and swabbed/tested positive
  Interventions: Other: NHANES smell and taste tests
- covid19 negative patients: participants who present with signs and symptoms suspected for covid19 and swabbed/tested negative
  Interventions: Other: NHANES smell and taste tests

INTERVENTIONS:
Other: NHANES smell and taste tests — participants will be asked to smell 8 cards of different odors and submit your choices in a given card, and so for 3 different taste tips (salty, bitter and neutral). participants will be asked to submit his choices in a given card as well. Then participants photograph those cards and send it via WhatsApp to a given number to be collected

SUMMARY:
COVID-19 has adversely affected the healthcare system across the world. The world was not prepared for global outbreak of infectious diseases. The rapid spread of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is enabling researchers worldwide to acquire a large amount of clinical data regarding coronavirus disease (COVID-19).

The COVID-19 infection severely affects the respiratory system in the critical cases and results in mortalities. The affected people experience a dry cough, fever, breathing problems, diarrhea, muscle pain, and sore throat. Besides that, some of the evidence from Italy, South Korea, China, and Spain suggest that the COVID-19 cases also lose their senses of smell and taste resulting in alterations in those patients.

The objective of this proposed study is to determine whether COVID-19 cases have Olfactory and gustatory dysfunctions as a hallmark indicator and can be used as diagnostic tools for the isolation of suspected people.

Investigators are presenting a prospective proportional case-control study that is conducted to investigate the COVID-19 cases with anosmia and /or Ageusia in a university hospital in Riyadh, Saudi Arabia. The sample size of this case series would be 250 cases of suspected COVID-19 patients. The cases included in the study are analyzed prospectively to determine if the cases had a history of anosmia and /or Ageusia, and then tested for the alteration of these senses through a panel of standardized odors/taste strips. That is looked at statistically allowing us to confirm the proposed effectiveness of these tests as a diagnostic tool.

DETAILED DESCRIPTION:
Upon identification of the patient in the triage area the research assistant will start the study by introducing the concept for the patient and then taking consent. The patient will go through the regular flow of patients in the ED and after being asked to do the swabs the research assistant will start the process of the study by testing the smell by the NHANES cards then directly assess the taste by the NHANES strips and documents the results on the cards and ask the patient to take a photo with his mobile and send it with his name to the primary investigator via a mobile application and dedicated phone number. The research assistant is the same person who is going to take the nasopharyngeal swab for the COVID-19 test. The cards are going to be collected in the negative pressure room of the patients and then discarded in the same room. The investigators in the study are not aware of which patient is answering what blinded investigator

Taste exam measures in NHANES The NHANES chemosensory tests used regional and whole mouth taste intensities of bitter and salt tastants as measures of taste function, which were similar to those implemented in the NIH Toolbox norming study. These NHANES taste measures were selected based on their ability to capture genetic and environmentally mediated variation in taste and for their potential relevance to diet and health.

Smell function in NHANES was assessed with an 8-item, odor identification test (Pocket Smell Tests™, Sensonics, Inc., Haddon Heights, NJ). Of many available psychophysical measures of olfactory function, odor identification tests are the most widely used in epidemiological and clinical settings, as they are quick, relatively inexpensive, and easy to administer. The odor identification test corresponds well with odor threshold tasks as well as other suprathreshold olfactory measures (e.g., discrimination, odor intensity), and hence is considered to be a rapid and accurate method for detecting olfactory dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1- Suspected cases of COVID -19 fulfilling the case definition of Saudi CDC 2- Adult patients

-

Exclusion Criteria:

1. The cases of children under the age of 12 years
2. Known patients with Kallmann's syndrome, CHARGE syndrome, Indifference to pain syndrome, ciliopathy disorders.
3. Known patient with congenital anomalies, absent smell sense, and absent taste sense.
4. Pregnant and lactating ladies
5. Patients with trigeminal nerve disease
6. Blind and deaf patients
7. Malingering.
8. Adults aged more than 65 years old.
9. Allergy to quinine products

   -

Ages: 12 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Upon identification of the patient in the triage area the research assistant will start the study by introducing the concept for the patient and then taking consent. The patient will go through the regular flow of patients in the ED and after being asked to do the swabs the research assistant will start the process of the study by testing the smell by the NHANES cards then directly assess the taste by the NHANES strips and documents the results on the cards
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
correlation of anosmia and ageusia to covid19 positive patients | from 1/06/2020 to 31/12/2020
  to how extent alteration of smell and taste senses is related to covid19 status

SECONDARY OUTCOMES:
objective assessment of severity of smell and taste senses alterations in covid19 patients | from 1/06/2020 to 31/12/2020
  to determine the range of sense affection ranging from total loss to mild form

CONTACTS AND LOCATIONS:
Overall Officials: OSAMA KENTAB, M.D, Principal Investigator — Princess Nourah Bint Abdulrahman University; AHMAD AALIBRAHIM, M.D, Study Director — Princess Nourah Bint Abdulrahman University; MARZOOQA ALENIZI, M.D, Study Chair — Princess Nourah Bint Abdulrahman University
Locations (2):
- Saudi Arabia (2):
  - Princess Nourah Bint Abdulrahman Univeristy, Riyadh, Central
  - prince Mohammed bin Abdulaziz Hospital, Riyadh, Central

IPD SHARING:
Plan to Share IPD: Undecided